CLINICAL TRIAL: NCT04627792
Title: Improving Child Mental Health Service Utilization in Ibadan Nigeria Using a Community Based Participatory Research Approach
Brief Title: Improving Child Mental Health Service Utilization in Ibadan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Howard University (Other)
Collaborators: University College Hospital, Ibadan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9414
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Waitlist Group (Other): We will use a switching replication design in which fifty guardians will be randomly assigned using a lottery to receive the intervention and fifty will be assigned to a group who will receive the intervention at a later time point
  Interventions: Behavioral: IUSECAMH Parent Intervention (Waitlist)

INTERVENTIONS:
Behavioral: IUSECAMH Parent Intervention (Waitlist) — We will use a switching replication design in which fifty guardians will be randomly assigned using a lottery to receive the intervention and fifty will be assigned to a group who will receive the intervention at a later time point

SUMMARY:
The investigators will develop and evaluate a community-based participatory intervention that will be principally guided by the model we test and confirm in Aim 1. To meet this second aim, ten guardian consultants will co-develop and co-implement a group intervention whose goal is to increase 100 guardians' recognition and knowledge of CAMH problems, perceived need for CAMH services, and willingness to use accessible services at UCH. The investigators will also evaluate the process of developing, planning, and administering a CBP intervention in Nigeria and draw broader implications for CBP programming in other LMICs.

DETAILED DESCRIPTION:
One hundred participants will be randomly recruited from the cohort of guardians who completed the interview in Phase 1 and expressed interest in participating in an intervention. The investigators will use a switching replication design in which fifty guardians will be randomly assigned using a lottery to receive the intervention and fifty will be assigned to a group who will receive the intervention at a later time point.127 The latter group will serve as a control in the first part of the intervention plan, and the roles will be switched in the second part. The investigators will initially propose 4 intervention sessions, each comprised of 2 meetings, lasting 1.5 hours each for 25 guardians. Two sessions will be conducted concurrently for Group 1 (n=50) followed by 2 sessions concurrently conducted for Group 2 (n=50). The program outcomes - guardian recognition and knowledge of CAMH problems, the perceived need for CAMH services, and willingness to use accessible CAMH services - will be measured with the same instruments administered in Aim 1

ELIGIBILITY:
Inclusion Criteria:

* Participated in Phase 1 of student (participated in structured interview)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Guardian recognition and knowledge of CAMH problems | up to 2 months
  This was assessed by the Yorùbá version of the Strengths and Difficulties Questionnaire - Parent Report (SDQ-P; Goodman, Ford, Simmons; Gatward, & Meltzer, 2000), a 25-item screening measure of emotional and behavioral problems for children aged 3 to 17-years extensively used in Africa (Hoosen et al., 2018). The SDQ-P utilized a three-point Likert scale (0=not true; 1=somewhat true; 2= certainly true). Five subscales were derived from the measure including conduct problems, inattention-hyperactivity, emotional symptoms, peer problems, and prosocial behavior. A total score was calculated by summing the subscales with higher scores indicating more recognition of CAMH problems (range= 0 - 50).
Perceived need for CAMH services | up to 2 months
  Adapted from the 2001 National Survey of Children with Special Health Care Needs in the United States (Porterfield & McBride, 2007), we asked caregivers: "Has there been a time in past year when your child/ any of your children (1) seemed sad and did not feel like doing anything over 2 weeks (yes/no)?; (2) not able to sit still or concentrate for long, always getting into trouble (yes/no)?; (3) displayed strange public behavior such as talking or laughing to themselves when no one is around (yes/no)?; (4) behaved in any way or reported feeling anyway that worried them, you, or others in your family or community?" If caregivers affirmed any of the 4 statements, they were subsequently asked: "During the past 12 months, was there any time when your child needed help because you were worried about the problems you just described? (yes/no)" Responses to the final question (0=no; 1=yes) was used to determine perceived need of CAMH services.
Willingness to use accessible CAMH services | up to 2 months
  Caregivers' willingness to use accessible mental health service was adapted from a study examining child mental health service utilization among parents in rural Appalachia (S. L. Williams & Polaha, 2014). Caregivers were asked "If my child experienced a mental health condition such as Dapo, Tola, and Moji [fictional characters with depression, ADHD, and psychosis in a previously administered section], I would take my child to see a healthcare provider at the mental health clinic for children and adolescents at UCH" (1 = Not at All, 6=Definitely).

CONTACTS AND LOCATIONS:
Overall Officials: Ezer Kang, Principal Investigator — Howard University

IPD SHARING:
Plan to Share IPD: No